CLINICAL TRIAL: NCT05702905
Title: Semaglutide Improves Metabolic Abnormalities and Fertility in Obese Infertile Women With Polycystic Ovary Syndrome: a Prospective, Randomized, Open, Controlled Study
Brief Title: Semaglutide Improves Metabolic Abnormalities and Fertility in Obese Infertile Women With Polycystic Ovary Syndrome
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Tingting ZHANG, Associate Chief Physician , Associate Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022CR04
Record Dates: First submitted 2022-12-23; First posted 2023-01-27 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: PCOS (Polycystic Ovary Syndrome); Semaglutide
Keywords: PCOS; semaglutide; obese; metabolic abnormality; fertility
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity | interventions — Metformin; semaglutide; Caloric Restriction; Exercise

STUDY DESIGN:
Intervention Model Description: All subjects will be randomized into three groups: metformin single, semaglutide single, both metformin and semaglutide.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- metformin (Active Comparator): About 25 subjects will be allocated to this group to receive metformin only, as the active comparator of semaglutide groups. Metformin used in this trial is Glucophage ( 500mg per tablet）produced by Bristol-Myers Squibb.The initial dose of metformin will be 500mg twice daily, which will be increased to 1000mg twice daily after two weeks, and then maintained until the end of treatment in total 12 weeks.
  Interventions: Drug: Metformin Hydrochloride 500 MG; Behavioral: calorie-restricted diet; Behavioral: physical exercise
- semaglutide (Experimental): About 25 subjects will be allocated to this group to receive semaglutide only, as one of the experimental groups. Semaglutide used in this trial is WEGOVY (semaglutide) injection produced by Novo Nordisk. Administer WEGOVY once weekly, on the same day each week, at any time of day, with or without meals. Inject subcutaneously in the abdomen, thigh or upper arm. Initiate at 0.25 mg once weekly for 4 weeks. In 4 week intervals, increase the dose until a dose of 1.0 mg is reached, and then maintained 1.0 mg until the end of treatment in total 12 weeks..
  Interventions: Drug: Semaglutide, 1.34 mg/mL; Behavioral: calorie-restricted diet; Behavioral: physical exercise
- semaglutide and metformin (Experimental): About 25 subjects will be allocated to this group to receive both semaglutide and metformin, as another of the experimental groups. Metformin used in this trial is Glucophage ( 500mg per tablet）produced by Bristol-Myers Squibb.The initial dose of metformin will be 500mg twice daily, which will be increased to 1000mg twice daily after two weeks, and then maintained until the end of treatment in total 12 weeks. Semaglutide used in this trial is WEGOVY (semaglutide) injection produced by Novo Nordisk. Administer WEGOVY once weekly, on the same day each week, at any time of day, with or without meals. Inject subcutaneously in the abdomen, thigh or upper arm. Initiate at 0.25 mg once weekly for 4 weeks. In 4 week intervals, increase the dose until a dose of 1.0 mg is reached, and then maintained 1.0 mg until the end of treatment in total 12 weeks.
  Interventions: Drug: Semaglutide, 1.34 mg/mL and Metformin Hydrochloride 500 MG; Behavioral: calorie-restricted diet; Behavioral: physical exercise

INTERVENTIONS:
Drug: Metformin Hydrochloride 500 MG — Metformin oral tablet (500mg per tablet) will be administered in a dose increasing mode: the initial dose will be 500mg twice daily, which will be increased to 1000mg twice daily after two weeks, and then maintained until the end of treatment in total 12 weeks.
  Other Names: Glucophage
  Arms: metformin
Drug: Semaglutide, 1.34 mg/mL — Inject semaglutide subcutaneously once weekly, on the same day each week, at any time of day, in a dose increasing mode: the initial dose of 0.25mg QW (once a week), increased to 0.5mg QW after 4 weeks, and increased to 1.0mg QW after another 4 weeks, and then maintained 1.0mg until the end of treatment in total 12 weeks.
  Other Names: WEGOVY
  Arms: semaglutide
Drug: Semaglutide, 1.34 mg/mL and Metformin Hydrochloride 500 MG — Both Semaglutide injection and Metformin oral tablet will be administered as described above.
  Other Names: WEGOVY and Glucophage
  Arms: semaglutide and metformin
Behavioral: calorie-restricted diet — All subjects after randomization will be reviewed and evaluated by a nutritionist, and then will receive diet guidance. The clinical nutritionist will develop a written nutrition plan for each subject. The nutrition plan of this study adopted the method of calorie restriction diet (CRD) to develop a diet, which required 83.68 kJ/kg of energy per day, 1.2 g/kg of protein per day, 40%~55% of carbohydrate energy supply ratio, and 20%~30% of fat energy supply ratio, to ensure the intake of vegetables, fruits and other rich dietary fiber, and drinking more than 1.5 L per day. The nutritionist will explain the method of food exchange in detail to enrich the food types of patients. The diet diary will be distributed to each subject, and the subjects will be required to make a return visit once every four weeks, return the diet diary each time, and receive guidance according to their compliance.
Behavioral: physical exercise — All subjects after randomization will be reviewed and evaluated by a trainer, and then will receive guidance of physical exercise.The trainer will formulate an exercise plan for each subject. The exercise plan consists of 30 minutes of moderate and low intensity continuous aerobic exercise every day, with a frequency of 5-7 days/week. The form of exercise can be determined according to personal hobbies, such as fast walking, jogging, climbing, swimming, etc. The exercise diary will be distributed to each subject, and the subjects are required to make a return visit once every four weeks, return the exercise diary each time, and the trainer will provide guidance to the subjects according to their compliance.

SUMMARY:
To investigate the efficacy of semaglutide in obese infertile women of childbearing age with polycystic ovary syndrome (PCOS), we design this prospective, randomized, open and controlled study. 75 obese infertile PCOS patients will be recruited and randomized into three groups: metformin, semaglutide and metformin+semaglutide, on the basis of calorie-restricted diet and physical exercise. All subjects will be treated for 12 weeks, and then stop taking the drug for at least 8 weeks to initiate ovulation induction or ovulation induction combined with artificial insemination. All subjects will be followed up for 24 weeks for pregnancy outcome. The primary endpoint of the study is the percentage of weight loss at 12 weeks of treatment. The secondary endpoints include HOMA-IR and androgen levels at 12 weeks of treatment, ovulation rate at 24 weeks of follow-up, clinical pregnancy rate and cumulative pregnancy rate, and depression, anxiety, diet and quality of life scores at 12 weeks of treatment.

DETAILED DESCRIPTION:
To investigate the efficacy of semaglutide in obese infertile women of childbearing age with polycystic ovary syndrome (PCOS), we design this prospective, randomized, open and controlled study. 75 obese infertile PCOS patients will be recruited and randomized into three groups: metformin, semaglutide and metformin+semaglutide, on the basis of calorie-restricted diet and physical exercise. Metformin and semaglutide will be administered in a dose increasing mode, and then maintain until the end of 12 weeks, and metabolic related indexes will be evaluated. After 12 weeks of treatment, all subjects will stop taking the drug for at least 8 weeks to initiate ovulation induction or ovulation induction combined with artificial insemination. All subjects will be followed up for 24 weeks to evaluate the fertility related indicators. The primary endpoint of the study is the percentage of weight loss at 12 weeks of treatment. The secondary endpoints include HOMA-IR and androgen levels at 12 weeks of treatment, ovulation rate at 24 weeks of follow-up, clinical pregnancy rate and cumulative pregnancy rate, and depression, anxiety, diet and quality of life scores at 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the PCOS diagnostic criteria (Rotterdam）
2. Age 22-40
3. BMI ≥ 28 kg/m2
4. Infertility: having normal sexual life and failing to conceive without contraception for more than 1 year
5. Willing to be pregnant, and her husband has no serious infertility

Exclusion Criteria:

1. History of acute pancreatitis, individual or family history of medullary thyroid cancer and multiple endocrine adenomas
2. Type 1 diabetes and special type diabetes
3. History of tumor
4. Serious cardiovascular and cerebrovascular disease, mental disease, liver or kidney disease
5. Metformin, GLP-1 RA and other drugs affecting reproductive and metabolic functions were used within 90 days before the study
6. Known allergy to metformin, GLP-1 RA and excipients
7. Severe endometriosis, low ovarian reserve, premature ovarian failure
8. Inability to tolerate pregnancy and ovulation induction therapy
9. Other conditions considered unsuitable for this study by researchers

Ages: 22 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 75 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage change in bodyweight at 12 weeks for semaglutide versus metformin | at the end of 12 weeks of treatment
  Difference between body weight at 12 weeks and baseline divided by baseline body weight
Achievement of weight reduction of at least 5% at 12 weeks for semaglutide versus metformin | at the end of 12 weeks of treatment
  Proportion of patients with weight loss at least 5% at 12 weeks of treatment

SECONDARY OUTCOMES:
HOMA-IR at 12 weeks of treatment | at the end of 12 weeks of treatment
  compare HOMA-IR at 12 weeks of treatment among three groups
testosterone level at 12 weeks of treatment | at the end of 12 weeks of treatment
  compare testosterone level at 12 weeks of treatment among three groups
androstenedione level at 12 weeks of treatment | at the end of 12 weeks of treatment
  compare androstenedione level at 12 weeks of treatment among three groups
FAI (Free Androgen Index) at 12 weeks of treatment | at the end of 12 weeks of treatment
  compare FAI at 12 weeks of treatment among three groups

OTHER OUTCOMES:
Depression score by self-rating depression scale (SDS）at 12 weeks of treatment | at the end of 12 weeks of treatment
  Zung self-rating depression scale (SDS) contains 20 items. Each item is divided into four grades according to the frequency of symptoms, of which 10 are positive and 10 are negative. Positive scoring question rated as 1, 2, 3 and 4 in turn and reverse scoring questions rated as 4, 3, 2 and 1. Add all the scores to get the total rough score, and then multiply the rough score by 1.25 to get the integral part as the standard score. The lower the score, the better. According to the criteria of Chinese population, the cut-off value of SDS standard score is 53 points, of which 53-62 points is mild depression, 63-72 points is moderate depression, and more than 73 points is severe depression. SDS standard score ≥ 50 indicates depressive symptoms. Depression severity is evaluated by cumulative score of each item/80. Those below 0.5 are not depressed; 0.5-0.59 is mild depression; 0.6-0.69 is moderate to severe; more than 0.7 is severe depression.
Anxiety score by self-rating anxiety scale (SAS）at 12 weeks of treatment | at the end of 12 weeks of treatment
  Zung self-reating anxiety scale (SAS) adopts a four-grade score, which is mainly used to assess the frequency of symptoms. The standard is: "1" means no or little time; "2" means sometimes; "3" means most of the time; "4" means most or all of the time. Of the 20 items, 15 items are stated in negative words, and scored in the order of 1-4 above. The remaining five items are stated in positive words and scored in reverse order of 4 to 1. The main statistical indicator of SAS is the total score. Add the scores of 20 items to get a rough score. Multiply the rough score by 1.25 and take the integer part to get the standard score. According to the criteria of Chinese population, the cut-off value of SAS standard score is 50 points, of which 50-59 points is mild anxiety, 60-69 points is moderate anxiety, and more than 70 points is severe anxiety.
Diet score by TFEQ-18 (three factor eating questionaire) at 12 weeks of treatment | at the end of 12 weeks of treatment
  The Three-Factor Eating Questionnaire Revised 18-item includes three dimensions of questions: non-controlled eating (9 items), cognitive restricted eating (6 items), and emotional eating (3 items). Uncontrolled eating refers to a tendency to lose control of excessive eating when feeling hungry or stimulated by external factors. Cognitive restriction refers to consciously limiting food intake to control weight or promote weight loss. Emotional eating refers to the tendency to overeat under some negative emotional conditions. Questions 1 to 18 are scored with 1 to 4 points. The total score of the three dimensions is the total score of the scale. The higher the score of each dimension of the questionnaire, the higher the tendency of uncontrolled eating, cognitive restriction of eating and emotional eating.
Quality of life score at 12 weeks of treatment | at the end of 12 weeks of treatment
  The World Health Organization Quality of Life (WHOQOL) - BREF can generate scores in four fields. The scale contains two independent analysis items: Q1 asks the individual's total subjective feelings about their own quality of life, and Q2 asks the individual's total subjective feelings about their own health status. The domain score is positive (that is, the higher the score, the better the quality of life). The domain score is obtained by calculating the average score of the items to which it belongs and multiplying by 4.
Ovulation rate at 24 weeks of follow-up after the end of treatment | at the end of 24 weeks of follow-up after the end of treatment
  Number of patients with ovulation after natural and ovulation induction treatment/total number of patients
Clinical pregnancy rate at 24 weeks of follow-up after the end of treatment | at the end of 24 weeks of follow-up after the end of treatment
  Clinical pregnancy rate=clinical pregnancy cycles/transplantation cycles
Cumulative pregnancy rate at 24 weeks of follow-up after the end of treatment | at the end of 24 weeks of follow-up after the end of treatment
  Cumulative pregnancy rate=number of all pregnant patients/total number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Tingting Zhang, M.D., Principal Investigator — Peking University First Hospital
Locations (1):
- PekingUFH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jensterle Sever M, Kocjan T, Pfeifer M, Kravos NA, Janez A. Short-term combined treatment with liraglutide and metformin leads to significant weight loss in obese women with polycystic ovary syndrome and previous poor response to metformin. Eur J Endocrinol. 2014 Feb 7;170(3):451-9. doi: 10.1530/EJE-13-0797. Print 2014 Mar. PMID 24362411
- [Result] Jensterle M, Kravos NA, Pfeifer M, Kocjan T, Janez A. A 12-week treatment with the long-acting glucagon-like peptide 1 receptor agonist liraglutide leads to significant weight loss in a subset of obese women with newly diagnosed polycystic ovary syndrome. Hormones (Athens). 2015 Jan-Mar;14(1):81-90. doi: 10.1007/BF03401383. PMID 25885106
- [Result] Salamun V, Jensterle M, Janez A, Vrtacnik Bokal E. Liraglutide increases IVF pregnancy rates in obese PCOS women with poor response to first-line reproductive treatments: a pilot randomized study. Eur J Endocrinol. 2018 Jul;179(1):1-11. doi: 10.1530/EJE-18-0175. Epub 2018 Apr 27. PMID 29703793
- [Result] Han Y, Li Y, He B. GLP-1 receptor agonists versus metformin in PCOS: a systematic review and meta-analysis. Reprod Biomed Online. 2019 Aug;39(2):332-342. doi: 10.1016/j.rbmo.2019.04.017. Epub 2019 Apr 25. PMID 31229399
- [Result] Cena H, Chiovato L, Nappi RE. Obesity, Polycystic Ovary Syndrome, and Infertility: A New Avenue for GLP-1 Receptor Agonists. J Clin Endocrinol Metab. 2020 Aug 1;105(8):e2695-709. doi: 10.1210/clinem/dgaa285. PMID 32442310
- [Result] Xing C, Zhao H, Zhang J, He B. Effect of metformin versus metformin plus liraglutide on gonadal and metabolic profiles in overweight patients with polycystic ovary syndrome. Front Endocrinol (Lausanne). 2022 Aug 17;13:945609. doi: 10.3389/fendo.2022.945609. eCollection 2022. PMID 36060969
- [Result] Papaetis GS, Kyriacou A. GLP-1 receptor agonists, polycystic ovary syndrome and reproductive dysfunction: Current research and future horizons. Adv Clin Exp Med. 2022 Nov;31(11):1265-1274. doi: 10.17219/acem/151695. PMID 35951627
- [Result] Ge JJ, Wang DJ, Song W, Shen SM, Ge WH. The effectiveness and safety of liraglutide in treating overweight/obese patients with polycystic ovary syndrome: a meta-analysis. J Endocrinol Invest. 2022 Feb;45(2):261-273. doi: 10.1007/s40618-021-01666-6. Epub 2021 Aug 29. PMID 34455568
- [Result] Liu X, Zhang Y, Zheng SY, Lin R, Xie YJ, Chen H, Zheng YX, Liu E, Chen L, Yan JH, Xu W, Mai TT, Gong Y. Efficacy of exenatide on weight loss, metabolic parameters and pregnancy in overweight/obese polycystic ovary syndrome. Clin Endocrinol (Oxf). 2017 Dec;87(6):767-774. doi: 10.1111/cen.13454. Epub 2017 Sep 13. PMID 28834553
- [Result] Ma RL, Deng Y, Wang YF, Zhu SY, Ding XS, Sun AJ. Short-term combined treatment with exenatide and metformin for overweight/obese women with polycystic ovary syndrome. Chin Med J (Engl). 2021 Nov 3;134(23):2882-2889. doi: 10.1097/CM9.0000000000001712. PMID 34732660
- [Result] Li R, Mai T, Zheng S, Zhang Y. Effect of metformin and exenatide on pregnancy rate and pregnancy outcomes in overweight or obese infertility PCOS women: long-term follow-up of an RCT. Arch Gynecol Obstet. 2022 Nov;306(5):1711-1721. doi: 10.1007/s00404-022-06700-3. Epub 2022 Jul 13. PMID 35829765

DOCUMENTS (2):
  • Study Protocol (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT05702905/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT05702905/SAP_001.pdf